CLINICAL TRIAL: NCT02507492
Title: RM-493 Treatment Trial in Proopiomelanocortin (POMC) Deficient Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, PD Dr. Susanna Wiegand, Principal Investigator, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RM-493-011; 2014-002392-28 (EudraCT Number)
Record Dates: First submitted 2015-05-29; First posted 2015-07-24 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Homozygous or Compound Heterozygous POMC, LEPR or PCSK1 Gene Mutation
Keywords: POMC, LEPR, PCSK1
MeSH Terms: interventions — setmelanotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RM-493 Once Daily (Experimental): Dose once daily in the morning
  Interventions: Drug: RM-493

INTERVENTIONS:
Drug: RM-493
  Other Names: setmelanotide

SUMMARY:
The purpose of this study is to evaluate the effects of a once daily subcutaneous (SC) injection of RM-493, in subjects with POMC (propiomelanocortin) or other related rare genetic mutations, on body weight, metabolic function and blood pressure. Patients who respond during the initial 84 days of treatment can enter into long-term (2-year) extensions. The study drug (RM-493) will be administered in an unblinded fashion.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Homozygous or compound heterozygous (different gene mutation on both alleles) POMC, LEPR or PCSK1 gene mutation
* Obesity (BMI > 30 kg/m2; + 2 BMI SDS)
* No other therapeutic option, which might cure the patient (e.g. bariatric surgery (see chapter 8))
* Negative Pregnancy test
* Highly effective contraception in women (defined as pearl index < 1), if necessary also for partners of test persons)
* No participation in other clinical trials according to AMG (Arzneimittelgesetz) (2 months before and after) at the time of this trial
* Normal or minimally elevated blood pressure (measured in 24RR monitoring or similar methods) according the guidelines of the ESH (European Society of Hypertension) and Deutsche Hochdruckliga: systolic > 159 mmHg/diastolic 99 mmHg
* sufficient kidney and liver function (Creatinine, ALT, AST)

  * normal values Alanine-Aminotransferase (ALT) (female): < 31 U/l
  * normal values Alanine-Aminotransferase (ALT) (male): < 41 U/l
  * normal values Aspartate-Aminotransferase (AST) (female > 17 years): < 35 U/l; (female < 17 years): 16- 46 U/l
  * normal values Aspartate-Aminotransferase (AST) (male > 17 years): < 50 U/l; (male < 17 years): 16-46 U/l
  * normal values bilirubins (male and female) up to 1,2 mg/dl
  * normal values Creatinine (female > 15 years): 0,51-0,95 mg/dl) ; (female < 15 years): 0,46-0,77 mg/dl
  * normal values Creatinine (male > 15 years): 0,67 - 1,17 mg/dl) ; (male < 15 years): 0,46-0,77 mg/dl

Exclusion Criteria:

* Pregnancy or Breastfeeding
* All contraindications against study medication (including auxiliary substances)
* Interactions with study medication
* Participation of the patient in a clinical study within the last 2 months
* Intolerance against albumin
* Concomitant diseases, impaired organ functions, except for known, concurrent GI disorders or other clinical findings expected in PCSK1 or LEPR gene disorders
* Renal insufficiency (Creatinine > 0,95 mg/dl (female), > 1,17 mg/dl (male))
* Impaired liver function (Bilirubins > 1.2 mg/dl)
* Neurological / psychiatric diseases
* HIV Infection
* Active Hepatitis B or C
* Melanoma or Melanoma occurrence in the family history
* Non-compliance
* Subjects who are legally detained in an official institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Effect of RM-493 on Body weight | Day 1 through Day 84
  Change of body weight after Treatment with RM-493.

SECONDARY OUTCOMES:
Effect of RM-493 on metabolic serum parameters | Day 1 through Day 84
  Measurement of the effect of RM-493 on metabolic serum parameters as measured by blood test.
Effect of RM-493 on blood pressure | Day 1 through Day 84
  Measurement of the effect of RM-493 on blood pressure by daily blood pressure measurements.
Effect of RM-493 on hunger | Day 1 through Day 84
  Measurement of the effect of RM-493 on hunger as measured by the Global Hunger Scale
Effect of RM-493 on body composition/Energy expenditure | Day 1 through Day 84
  Measurement of the effect of RM-493 on body composition/Energy expenditure
Effect of RM-493 on weight loss after treatment continuation of 2 years | Day 1 through Day 730
  Measurement of the effect of RM-493 on weight loss after treatment continuation of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany